CLINICAL TRIAL: NCT01298648
Title: Special Investigation (All Cases Investigation in Patients With Crohn's Disease)
Brief Title: Special Investigation in Patients With Crohn's Disease (All Patients Investigation)
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-706
Record Dates: First submitted 2011-01-26; First posted 2011-02-18 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2014-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Humira: Participants who were prescribed Humira per approved prescribing information of Humira in Japan.

SUMMARY:
This study will be conducted to assess adverse drug reactions, incidence of adverse events, and factors that may affect the safety and effectiveness of Humira for the treatment of Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients with moderate or severe active Crohn's disease who are not responding well to conventional therapy and receive Humira will be enrolled in the survey

Exclusion Criteria:

Contraindications according to the Package Insert

* Patients who have serious infections
* Patients who have tuberculosis
* Patients with a history of hypersensitivity to any ingredient of Humira
* Patients who have demyelinating disease or with a history of demyelinating disease
* Patients who have congestive cardiac failure

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who receive Humira for the treatment of Crohn's Disease
Sampling Method: Non-Probability Sample
Enrollment: 1716 (Actual)
Dates: Start 2010-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sadanori Abe, Study Director — AbbVie
Locations (1131):
- Japan (1131):
  - Site Reference ID/Investigator# 60378, Abiko
  - Site Reference ID/Investigator# 48682, Aichi
  - Site Reference ID/Investigator# 48693, Aichi
  - Site Reference ID/Investigator# 49011, Aichi
  - Site Reference ID/Investigator# 49013, Aichi
  - Site Reference ID/Investigator# 49015, Aichi
  - Site Reference ID/Investigator# 49016, Aichi
  - Site Reference ID/Investigator# 49019, Aichi
  - Site Reference ID/Investigator# 55615, Aichi
  - Site Reference ID/Investigator# 55616, Aichi
  - Site Reference ID/Investigator# 55865, Aichi
  - Site Reference ID/Investigator# 55869, Aichi
  - Site Reference ID/Investigator# 55870, Aichi
  - Site Reference ID/Investigator# 55871, Aichi
  - Site Reference ID/Investigator# 55872, Aichi
  - Site Reference ID/Investigator# 55873, Aichi
  - Site Reference ID/Investigator# 55874, Aichi
  - Site Reference ID/Investigator# 55875, Aichi
  - Site Reference ID/Investigator# 55876, Aichi
  - Site Reference ID/Investigator# 55877, Aichi
  - Site Reference ID/Investigator# 60203, Aichi
  - Site Reference ID/Investigator# 60205, Aichi
  - Site Reference ID/Investigator# 60244, Aichi
  - Site Reference ID/Investigator# 60508, Aichi
  - Site Reference ID/Investigator# 65148, Aichi
  - Site Reference ID/Investigator# 67162, Aichi
  - Site Reference ID/Investigator# 48652, Aizu-Wakamatsu
  - Site Reference ID/Investigator# 55758, Akashi
  - Site Reference ID/Investigator# 89873, Akashi
  - Site Reference ID/Investigator# 60398, Aki-gun, Hiroshima
  - Site Reference ID/Investigator# 60401, Aki-gun, Hiroshima
  - Site Reference ID/Investigator# 48650, Akita
  - Site Reference ID/Investigator# 55660, Akita
  - Site Reference ID/Investigator# 55705, Akita
  - Site Reference ID/Investigator# 55905, Akita
  - Site Reference ID/Investigator# 55906, Akita
  - Site Reference ID/Investigator# 55907, Akita
  - Site Reference ID/Investigator# 55909, Akita
  - Site Reference ID/Investigator# 60190, Akita
  - Site Reference ID/Investigator# 60261, Akita
  - Site Reference ID/Investigator# 60376, Akita
  - Site Reference ID/Investigator# 55742, Amagasaki
  - Site Reference ID/Investigator# 56030, Anan
  - Site Reference ID/Investigator# 49026, Anjo
  - Site Reference ID/Investigator# 55617, Anjo
  - Site Reference ID/Investigator# 48797, Aomori
  - Site Reference ID/Investigator# 55584, Aomori
  - Site Reference ID/Investigator# 55585, Aomori
  - Site Reference ID/Investigator# 55897, Aomori
  - Site Reference ID/Investigator# 55898, Aomori
  - Site Reference ID/Investigator# 55899, Aomori
  - Site Reference ID/Investigator# 55900, Aomori
  - Site Reference ID/Investigator# 60509, Aomori
  - Site Reference ID/Investigator# 65111, Aomori
  - Site Reference ID/Investigator# 65144, Aomori
  - Site Reference ID/Investigator# 80014, Aomori
  - Site Reference ID/Investigator# 48648, Asahikawa
  - Site Reference ID/Investigator# 55797, Asahikawa
  - Site Reference ID/Investigator# 56032, Awa
  - Site Reference ID/Investigator# 55778, Ayabe
  - Site Reference ID/Investigator# 80233, Azumino
  - Site Reference ID/Investigator# 80220, Beppu
  - Site Reference ID/Investigator# 48668, Chiba
  - Site Reference ID/Investigator# 48672, Chiba
  - Site Reference ID/Investigator# 49000, Chiba
  - Site Reference ID/Investigator# 49002, Chiba
  - Site Reference ID/Investigator# 49006, Chiba
  - Site Reference ID/Investigator# 55647, Chiba
  - Site Reference ID/Investigator# 55796, Chiba
  - Site Reference ID/Investigator# 55820, Chiba
  - Site Reference ID/Investigator# 55821, Chiba
  - Site Reference ID/Investigator# 55822, Chiba
  - Site Reference ID/Investigator# 55826, Chiba
  - Site Reference ID/Investigator# 55827, Chiba
  - Site Reference ID/Investigator# 55841, Chiba
  - Site Reference ID/Investigator# 60257, Chiba
  - Site Reference ID/Investigator# 65115, Chiba
  - Site Reference ID/Investigator# 65116, Chiba
  - Site Reference ID/Investigator# 65117, Chiba
  - Site Reference ID/Investigator# 65138, Chiba
  - Site Reference ID/Investigator# 67169, Chiba
  - Site Reference ID/Investigator# 79900, Chiba
  - Site Reference ID/Investigator# 89820, Chichibu
  - Site Reference ID/Investigator# 49074, Chikushino-shi
  - Site Reference ID/Investigator# 55880, Chita
  - Site Reference ID/Investigator# 60210, Chita
  - Site Reference ID/Investigator# 55886, Chitose
  - Site Reference ID/Investigator# 55920, Chūō
  - Site Reference ID/Investigator# 80236, Ebetsu
  - Site Reference ID/Investigator# 49076, Ehime
  - Site Reference ID/Investigator# 55583, Ehime
  - Site Reference ID/Investigator# 56026, Ehime
  - Site Reference ID/Investigator# 56044, Ehime
  - Site Reference ID/Investigator# 65155, Ehime
  - Site Reference ID/Investigator# 79935, Esashi
  - Site Reference ID/Investigator# 89827, Fuji
  - Site Reference ID/Investigator# 48688, Fujieda
  - Site Reference ID/Investigator# 48689, Fujinomiya
  - Site Reference ID/Investigator# 79876, Fujisawa
  - Site Reference ID/Investigator# 48744, Fukui
  - Site Reference ID/Investigator# 55190, Fukui
  - Site Reference ID/Investigator# 55312, Fukui
  - Site Reference ID/Investigator# 55771, Fukui
  - Site Reference ID/Investigator# 55793, Fukui
  - Site Reference ID/Investigator# 80234, Fukui
  - Site Reference ID/Investigator# 48760, Fukuoka
  - Site Reference ID/Investigator# 48761, Fukuoka
  - Site Reference ID/Investigator# 48762, Fukuoka
  - Site Reference ID/Investigator# 48763, Fukuoka
  - Site Reference ID/Investigator# 48764, Fukuoka
  - Site Reference ID/Investigator# 48767, Fukuoka
  - Site Reference ID/Investigator# 48784, Fukuoka
  - Site Reference ID/Investigator# 49069, Fukuoka
  - Site Reference ID/Investigator# 49080, Fukuoka
  - Site Reference ID/Investigator# 49083, Fukuoka
  - Site Reference ID/Investigator# 49084, Fukuoka
  - Site Reference ID/Investigator# 49086, Fukuoka
  - Site Reference ID/Investigator# 55305, Fukuoka
  - Site Reference ID/Investigator# 56036, Fukuoka
  - Site Reference ID/Investigator# 56037, Fukuoka
  - Site Reference ID/Investigator# 56040, Fukuoka
  - Site Reference ID/Investigator# 56041, Fukuoka
  - Site Reference ID/Investigator# 56042, Fukuoka
  - Site Reference ID/Investigator# 56043, Fukuoka
  - Site Reference ID/Investigator# 56048, Fukuoka
  - Site Reference ID/Investigator# 56052, Fukuoka
  - Site Reference ID/Investigator# 60426, Fukuoka
  - Site Reference ID/Investigator# 60530, Fukuoka
  - Site Reference ID/Investigator# 60558, Fukuoka
  - Site Reference ID/Investigator# 65130, Fukuoka
  - Site Reference ID/Investigator# 65131, Fukuoka
  - Site Reference ID/Investigator# 65146, Fukuoka
  - Site Reference ID/Investigator# 65151, Fukuoka
  - Site Reference ID/Investigator# 68637, Fukuoka
  - Site Reference ID/Investigator# 68638, Fukuoka
  - Site Reference ID/Investigator# 90413, Fukuoka
  - Site Reference ID/Investigator# 48984, Fukushima
  - Site Reference ID/Investigator# 55163, Fukushima
  - Site Reference ID/Investigator# 55316, Fukushima
  - Site Reference ID/Investigator# 55597, Fukushima
  - Site Reference ID/Investigator# 55720, Fukushima
  - Site Reference ID/Investigator# 55798, Fukushima
  - Site Reference ID/Investigator# 55947, Fukushima
  - Site Reference ID/Investigator# 55948, Fukushima
  - Site Reference ID/Investigator# 55949, Fukushima
  - Site Reference ID/Investigator# 55950, Fukushima
  - Site Reference ID/Investigator# 55951, Fukushima
  - Site Reference ID/Investigator# 60196, Fukushima
  - Site Reference ID/Investigator# 60248, Fukushima
  - Site Reference ID/Investigator# 60386, Fukushima
  - Site Reference ID/Investigator# 60563, Fukushima
  - Site Reference ID/Investigator# 90396, Fukushima
  - Site Reference ID/Investigator# 55789, Fukuyama
  - Site Reference ID/Investigator# 56000, Fukuyama
  - Site Reference ID/Investigator# 90416, Fukuyama
  - Site Reference ID/Investigator# 48697, Gifu
  - Site Reference ID/Investigator# 49020, Gifu
  - Site Reference ID/Investigator# 49022, Gifu
  - Site Reference ID/Investigator# 55319, Gifu
  - Site Reference ID/Investigator# 55620, Gifu
  - Site Reference ID/Investigator# 55621, Gifu
  - Site Reference ID/Investigator# 55624, Gifu
  - Site Reference ID/Investigator# 55626, Gifu
  - Site Reference ID/Investigator# 55627, Gifu
  - Site Reference ID/Investigator# 55629, Gifu
  - Site Reference ID/Investigator# 60246, Gifu
  - Site Reference ID/Investigator# 60258, Gifu
  - Site Reference ID/Investigator# 60262, Gifu
  - Site Reference ID/Investigator# 60368, Gifu
  - Site Reference ID/Investigator# 60387, Gifu
  - Site Reference ID/Investigator# 60412, Gifu
  - Site Reference ID/Investigator# 60423, Gifu
  - Site Reference ID/Investigator# 60556, Gifu
  - Site Reference ID/Investigator# 60559, Gifu
  - Site Reference ID/Investigator# 67159, Gifu
  - Site Reference ID/Investigator# 48998, Gunma
  - Site Reference ID/Investigator# 55965, Gunma
  - Site Reference ID/Investigator# 55966, Gunma
  - Site Reference ID/Investigator# 55968, Gunma
  - Site Reference ID/Investigator# 60192, Gunma
  - Site Reference ID/Investigator# 60214, Gunma
  - Site Reference ID/Investigator# 60380, Gunma
  - Site Reference ID/Investigator# 65105, Gunma
  - Site Reference ID/Investigator# 67157, Gunma
  - Site Reference ID/Investigator# 67158, Gunma
  - Site Reference ID/Investigator# 55902, Hachinohe
  - Site Reference ID/Investigator# 60363, Hachinohe
  - Site Reference ID/Investigator# 48646, Hakodate
  - Site Reference ID/Investigator# 89856, Hakodate
  - Site Reference ID/Investigator# 48690, Hamamatsu
  - Site Reference ID/Investigator# 48691, Hamamatsu
  - Site Reference ID/Investigator# 55317, Hamamatsu
  - Site Reference ID/Investigator# 55613, Hamamatsu
  - Site Reference ID/Investigator# 55790, Hamamatsu
  - Site Reference ID/Investigator# 89817, Hamamatsu
  - Site Reference ID/Investigator# 55622, Hashima
  - Site Reference ID/Investigator# 55623, Hashima
  - Site Reference ID/Investigator# 56001, Higashihiroshima
  - Site Reference ID/Investigator# 55794, Higashiosaka
  - Site Reference ID/Investigator# 71467, Higashiosaka
  - Site Reference ID/Investigator# 55593, Himeji
  - Site Reference ID/Investigator# 55599, Himeji
  - Site Reference ID/Investigator# 55703, Himeji
  - Site Reference ID/Investigator# 90401, Himeji
  - Site Reference ID/Investigator# 55650, Hirakata
  - Site Reference ID/Investigator# 55311, Hirosaki
  - Site Reference ID/Investigator# 89813, Hirosaki
  - Site Reference ID/Investigator# 48751, Hiroshima
  - Site Reference ID/Investigator# 49063, Hiroshima
  - Site Reference ID/Investigator# 49064, Hiroshima
  - Site Reference ID/Investigator# 49068, Hiroshima
  - Site Reference ID/Investigator# 55164, Hiroshima
  - Site Reference ID/Investigator# 55574, Hiroshima
  - Site Reference ID/Investigator# 55581, Hiroshima
  - Site Reference ID/Investigator# 55601, Hiroshima
  - Site Reference ID/Investigator# 55694, Hiroshima
  - Site Reference ID/Investigator# 55997, Hiroshima
  - Site Reference ID/Investigator# 56002, Hiroshima
  - Site Reference ID/Investigator# 56003, Hiroshima
  - Site Reference ID/Investigator# 56004, Hiroshima
  - Site Reference ID/Investigator# 56005, Hiroshima
  - Site Reference ID/Investigator# 56007, Hiroshima
  - Site Reference ID/Investigator# 56008, Hiroshima
  - Site Reference ID/Investigator# 56010, Hiroshima
  - Site Reference ID/Investigator# 56014, Hiroshima
  - Site Reference ID/Investigator# 60554, Hiroshima
  - Site Reference ID/Investigator# 60560, Hiroshima
  - Site Reference ID/Investigator# 55588, Hitachi
  - Site Reference ID/Investigator# 56068, Hitoyoshi
  - Site Reference ID/Investigator# 48643, Hokkaido
  - Site Reference ID/Investigator# 48644, Hokkaido
  - Site Reference ID/Investigator# 48645, Hokkaido
  - Site Reference ID/Investigator# 48788, Hokkaido
  - Site Reference ID/Investigator# 48792, Hokkaido
  - Site Reference ID/Investigator# 48793, Hokkaido
  - Site Reference ID/Investigator# 48795, Hokkaido
  - Site Reference ID/Investigator# 48796, Hokkaido
  - Site Reference ID/Investigator# 55315, Hokkaido
  - Site Reference ID/Investigator# 55785, Hokkaido
  - Site Reference ID/Investigator# 55791, Hokkaido
  - Site Reference ID/Investigator# 55804, Hokkaido
  - Site Reference ID/Investigator# 55878, Hokkaido
  - Site Reference ID/Investigator# 55885, Hokkaido
  - Site Reference ID/Investigator# 55887, Hokkaido
  - Site Reference ID/Investigator# 55888, Hokkaido
  - Site Reference ID/Investigator# 55889, Hokkaido
  - Site Reference ID/Investigator# 55891, Hokkaido
  - Site Reference ID/Investigator# 55892, Hokkaido
  - Site Reference ID/Investigator# 55893, Hokkaido
  - Site Reference ID/Investigator# 55894, Hokkaido
  - Site Reference ID/Investigator# 55895, Hokkaido
  - Site Reference ID/Investigator# 60193, Hokkaido
  - Site Reference ID/Investigator# 60201, Hokkaido
  - Site Reference ID/Investigator# 60540, Hokkaido
  - Site Reference ID/Investigator# 60552, Hokkaido
  - Site Reference ID/Investigator# 60557, Hokkaido
  - Site Reference ID/Investigator# 65109, Hokkaido
  - Site Reference ID/Investigator# 65110, Hokkaido
  - Site Reference ID/Investigator# 48755, Houfu
  - Site Reference ID/Investigator# 80219, Houfu
  - Site Reference ID/Investigator# 48707, Hyōgo
  - Site Reference ID/Investigator# 48708, Hyōgo
  - Site Reference ID/Investigator# 48710, Hyōgo
  - Site Reference ID/Investigator# 48712, Hyōgo
  - Site Reference ID/Investigator# 48713, Hyōgo
  - Site Reference ID/Investigator# 49042, Hyōgo
  - Site Reference ID/Investigator# 49046, Hyōgo
  - Site Reference ID/Investigator# 49047, Hyōgo
  - Site Reference ID/Investigator# 55156, Hyōgo
  - Site Reference ID/Investigator# 55691, Hyōgo
  - Site Reference ID/Investigator# 55743, Hyōgo
  - Site Reference ID/Investigator# 55744, Hyōgo
  - Site Reference ID/Investigator# 55746, Hyōgo
  - Site Reference ID/Investigator# 55748, Hyōgo
  - Site Reference ID/Investigator# 55749, Hyōgo
  - Site Reference ID/Investigator# 55750, Hyōgo
  - Site Reference ID/Investigator# 55752, Hyōgo
  - Site Reference ID/Investigator# 55753, Hyōgo
  - Site Reference ID/Investigator# 55755, Hyōgo
  - Site Reference ID/Investigator# 55756, Hyōgo
  - Site Reference ID/Investigator# 55757, Hyōgo
  - Site Reference ID/Investigator# 55759, Hyōgo
  - Site Reference ID/Investigator# 60215, Hyōgo
  - Site Reference ID/Investigator# 60224, Hyōgo
  - Site Reference ID/Investigator# 60251, Hyōgo
  - Site Reference ID/Investigator# 60364, Hyōgo
  - Site Reference ID/Investigator# 60388, Hyōgo
  - Site Reference ID/Investigator# 60389, Hyōgo
  - Site Reference ID/Investigator# 60402, Hyōgo
  - Site Reference ID/Investigator# 60528, Hyōgo
  - Site Reference ID/Investigator# 60531, Hyōgo
  - Site Reference ID/Investigator# 65143, Hyōgo
  - Site Reference ID/Investigator# 68641, Hyōgo
  - Site Reference ID/Investigator# 48994, Ibaraki
  - Site Reference ID/Investigator# 49008, Ibaraki
  - Site Reference ID/Investigator# 55596, Ibaraki
  - Site Reference ID/Investigator# 55693, Ibaraki
  - Site Reference ID/Investigator# 55955, Ibaraki
  - Site Reference ID/Investigator# 55957, Ibaraki
  - Site Reference ID/Investigator# 55958, Ibaraki
  - Site Reference ID/Investigator# 55959, Ibaraki
  - Site Reference ID/Investigator# 60253, Ibaraki
  - Site Reference ID/Investigator# 60362, Ibaraki
  - Site Reference ID/Investigator# 60407, Ibaraki
  - Site Reference ID/Investigator# 60524, Ibaraki
  - Site Reference ID/Investigator# 48991, Ibaraki-ken
  - Site Reference ID/Investigator# 55824, Ichihara
  - Site Reference ID/Investigator# 55825, Ichihara
  - Site Reference ID/Investigator# 48667, Ichikawa
  - Site Reference ID/Investigator# 60513, Ichinomiya
  - Site Reference ID/Investigator# 60216, Ichinoseki
  - Site Reference ID/Investigator# 90415, Ichinoseki
  - Site Reference ID/Investigator# 67156, Iijima
  - Site Reference ID/Investigator# 49078, Iizuka
  - Site Reference ID/Investigator# 55685, Ikoma
  - Site Reference ID/Investigator# 49043, Ikomo, Nara
  - Site Reference ID/Investigator# 55313, Imabari
  - Site Reference ID/Investigator# 80222, Ina
  - Site Reference ID/Investigator# 55704, Inashiki
  - Site Reference ID/Investigator# 94893, Inazawa
  - Site Reference ID/Investigator# 60510, Inzai
  - Site Reference ID/Investigator# 94804, Isa
  - Site Reference ID/Investigator# 94805, Isa
  - Site Reference ID/Investigator# 55571, Isehara
  - Site Reference ID/Investigator# 48657, Isesaki
  - Site Reference ID/Investigator# 49052, Ishikawa
  - Site Reference ID/Investigator# 55162, Ishikawa
  - Site Reference ID/Investigator# 55765, Ishikawa
  - Site Reference ID/Investigator# 55767, Ishikawa
  - Site Reference ID/Investigator# 55768, Ishikawa
  - Site Reference ID/Investigator# 55769, Ishikawa
  - Site Reference ID/Investigator# 55770, Ishikawa
  - Site Reference ID/Investigator# 60555, Ishikawa
  - Site Reference ID/Investigator# 65125, Ishikawa
  - Site Reference ID/Investigator# 65126, Ishikawa
  - Site Reference ID/Investigator# 60375, Itami
  - Site Reference ID/Investigator# 55946, Iwaki
  - Site Reference ID/Investigator# 49060, Iwakuni
  - Site Reference ID/Investigator# 55612, Iwata
  - Site Reference ID/Investigator# 49048, Izumiōtsu
  - Site Reference ID/Investigator# 55673, Izumisano
  - Site Reference ID/Investigator# 49061, Izumo
  - Site Reference ID/Investigator# 49062, Izumo
  - Site Reference ID/Investigator# 55882, Izunokuni
  - Site Reference ID/Investigator# 84095, Izunokuni
  - Site Reference ID/Investigator# 55954, Jōetsu
  - Site Reference ID/Investigator# 79878, Jyoyo
  - Site Reference ID/Investigator# 49070, Kagawa
  - Site Reference ID/Investigator# 55716, Kagawa
  - Site Reference ID/Investigator# 55782, Kagawa
  - Site Reference ID/Investigator# 55805, Kagawa
  - Site Reference ID/Investigator# 56017, Kagawa
  - Site Reference ID/Investigator# 56018, Kagawa
  - Site Reference ID/Investigator# 56019, Kagawa
  - Site Reference ID/Investigator# 56020, Kagawa
  - Site Reference ID/Investigator# 56021, Kagawa
  - Site Reference ID/Investigator# 56022, Kagawa
  - Site Reference ID/Investigator# 56025, Kagawa
  - Site Reference ID/Investigator# 60221, Kagawa
  - Site Reference ID/Investigator# 65129, Kagawa
  - Site Reference ID/Investigator# 48777, Kagoshima
  - Site Reference ID/Investigator# 48778, Kagoshima
  - Site Reference ID/Investigator# 48779, Kagoshima
  - Site Reference ID/Investigator# 49091, Kagoshima
  - Site Reference ID/Investigator# 49092, Kagoshima
  - Site Reference ID/Investigator# 56069, Kagoshima
  - Site Reference ID/Investigator# 56070, Kagoshima
  - Site Reference ID/Investigator# 56077, Kagoshima
  - Site Reference ID/Investigator# 56079, Kagoshima
  - Site Reference ID/Investigator# 60222, Kagoshima
  - Site Reference ID/Investigator# 60377, Kagoshima
  - Site Reference ID/Investigator# 60517, Kagoshima
  - Site Reference ID/Investigator# 65134, Kagoshima
  - Site Reference ID/Investigator# 65135, Kagoshima
  - Site Reference ID/Investigator# 94802, Kagoshima
  - Site Reference ID/Investigator# 65122, Kaizuka
  - Site Reference ID/Investigator# 55625, Kakamigahara
  - Site Reference ID/Investigator# 89831, Kako
  - Site Reference ID/Investigator# 48680, Kamakura
  - Site Reference ID/Investigator# 84098, Kamo
  - Site Reference ID/Investigator# 49001, Kamogawa
  - Site Reference ID/Investigator# 55663, Kanagawa
  - Site Reference ID/Investigator# 55699, Kanagawa
  - Site Reference ID/Investigator# 55802, Kanagawa
  - Site Reference ID/Investigator# 55850, Kanagawa
  - Site Reference ID/Investigator# 55857, Kanagawa
  - Site Reference ID/Investigator# 55859, Kanagawa
  - Site Reference ID/Investigator# 55860, Kanagawa
  - Site Reference ID/Investigator# 55861, Kanagawa
  - Site Reference ID/Investigator# 55862, Kanagawa
  - Site Reference ID/Investigator# 55863, Kanagawa
  - Site Reference ID/Investigator# 55864, Kanagawa
  - Site Reference ID/Investigator# 60415, Kanagawa
  - Site Reference ID/Investigator# 60416, Kanagawa
  - Site Reference ID/Investigator# 60422, Kanagawa
  - Site Reference ID/Investigator# 60504, Kanagawa
  - Site Reference ID/Investigator# 60518, Kanagawa
  - Site Reference ID/Investigator# 60520, Kanagawa
  - Site Reference ID/Investigator# 60521, Kanagawa
  - Site Reference ID/Investigator# 60566, Kanagawa
  - Site Reference ID/Investigator# 55194, Kanazawa
  - Site Reference ID/Investigator# 55600, Kanazawa
  - Site Reference ID/Investigator# 55763, Kanazawa
  - Site Reference ID/Investigator# 55764, Kanazawa
  - Site Reference ID/Investigator# 55853, Kanazawa
  - Site Reference ID/Investigator# 79877, Kanazawa
  - Site Reference ID/Investigator# 84093, Kanazawa
  - Site Reference ID/Investigator# 48695, Kariya
  - Site Reference ID/Investigator# 55189, Kashihara
  - Site Reference ID/Investigator# 55602, Kashihara
  - Site Reference ID/Investigator# 48671, Kashiwa
  - Site Reference ID/Investigator# 84114, Kasukabe
  - Site Reference ID/Investigator# 84116, Kawachi-Nagano
  - Site Reference ID/Investigator# 48704, Kawachinago
  - Site Reference ID/Investigator# 48675, Kawagoe
  - Site Reference ID/Investigator# 55844, Kawagoe
  - Site Reference ID/Investigator# 67154, Kawagoe
  - Site Reference ID/Investigator# 60523, Kawanishi
  - Site Reference ID/Investigator# 55324, Kawasaki
  - Site Reference ID/Investigator# 55843, Kawasaki
  - Site Reference ID/Investigator# 55851, Kawasaki
  - Site Reference ID/Investigator# 60533, Kawasaki
  - Site Reference ID/Investigator# 60542, Kawasaki
  - Site Reference ID/Investigator# 79953, Kawasaki
  - Site Reference ID/Investigator# 55614, Kikukawa
  - Site Reference ID/Investigator# 49095, Kirishima
  - Site Reference ID/Investigator# 55823, Kisarazu
  - Site Reference ID/Investigator# 48765, Kitakyushu
  - Site Reference ID/Investigator# 49077, Kitakyushu
  - Site Reference ID/Investigator# 49079, Kitakyushu
  - Site Reference ID/Investigator# 49081, Kitakyushu
  - Site Reference ID/Investigator# 55618, Kitakyushu
  - Site Reference ID/Investigator# 56039, Kitakyushu
  - Site Reference ID/Investigator# 60519, Kitakyushu
  - Site Reference ID/Investigator# 60537, Kitakyushu
  - Site Reference ID/Investigator# 71473, Kitakyushu
  - Site Reference ID/Investigator# 48709, Kobe
  - Site Reference ID/Investigator# 55157, Kobe
  - Site Reference ID/Investigator# 55573, Kobe
  - Site Reference ID/Investigator# 55692, Kobe
  - Site Reference ID/Investigator# 55745, Kobe
  - Site Reference ID/Investigator# 55747, Kobe
  - Site Reference ID/Investigator# 55751, Kobe
  - Site Reference ID/Investigator# 48759, Kochi
  - Site Reference ID/Investigator# 49072, Kochi
  - Site Reference ID/Investigator# 55657, Kochi
  - Site Reference ID/Investigator# 55719, Kochi
  - Site Reference ID/Investigator# 56027, Kochi
  - Site Reference ID/Investigator# 56031, Kochi
  - Site Reference ID/Investigator# 56033, Kochi
  - Site Reference ID/Investigator# 56034, Kochi
  - Site Reference ID/Investigator# 60195, Kochi
  - Site Reference ID/Investigator# 60260, Kochi
  - Site Reference ID/Investigator# 60264, Kochi
  - Site Reference ID/Investigator# 60408, Kochi
  - Site Reference ID/Investigator# 55969, Kofu
  - Site Reference ID/Investigator# 79875, Kofu
  - Site Reference ID/Investigator# 48995, Koga
  - Site Reference ID/Investigator# 55924, Komagane
  - Site Reference ID/Investigator# 84097, Komaki
  - Site Reference ID/Investigator# 55766, Komatsu
  - Site Reference ID/Investigator# 49017, Koshigaya
  - Site Reference ID/Investigator# 94800, Koshigaya
  - Site Reference ID/Investigator# 55307, Kōnan
  - Site Reference ID/Investigator# 48654, Kōriyama
  - Site Reference ID/Investigator# 55603, Kōriyama
  - Site Reference ID/Investigator# 67265, Kōriyama
  - Site Reference ID/Investigator# 80013, Kōriyama
  - Site Reference ID/Investigator# 56016, Kudamatsu
  - Site Reference ID/Investigator# 55904, Kuji
  - Site Reference ID/Investigator# 48773, Kumamoto
  - Site Reference ID/Investigator# 48774, Kumamoto
  - Site Reference ID/Investigator# 48775, Kumamoto
  - Site Reference ID/Investigator# 48776, Kumamoto
  - Site Reference ID/Investigator# 48781, Kumamoto
  - Site Reference ID/Investigator# 49094, Kumamoto
  - Site Reference ID/Investigator# 56065, Kumamoto
  - Site Reference ID/Investigator# 56066, Kumamoto
  - Site Reference ID/Investigator# 56067, Kumamoto
  - Site Reference ID/Investigator# 56071, Kumamoto
  - Site Reference ID/Investigator# 60220, Kumamoto
  - Site Reference ID/Investigator# 60367, Kumamoto
  - Site Reference ID/Investigator# 60369, Kumamoto
  - Site Reference ID/Investigator# 60382, Kumamoto
  - Site Reference ID/Investigator# 60385, Kumamoto
  - Site Reference ID/Investigator# 60411, Kumamoto
  - Site Reference ID/Investigator# 60427, Kumamoto
  - Site Reference ID/Investigator# 60550, Kumamoto
  - Site Reference ID/Investigator# 65141, Kumamoto
  - Site Reference ID/Investigator# 79894, Kumamoto
  - Site Reference ID/Investigator# 79897, Kumamoto
  - Site Reference ID/Investigator# 84113, Kumamoto
  - Site Reference ID/Investigator# 48748, Kurashiki
  - Site Reference ID/Investigator# 55169, Kurashiki
  - Site Reference ID/Investigator# 67165, Kurashiki
  - Site Reference ID/Investigator# 56006, Kure
  - Site Reference ID/Investigator# 55761, Kurobe
  - Site Reference ID/Investigator# 48766, Kurume
  - Site Reference ID/Investigator# 48768, Kurume
  - Site Reference ID/Investigator# 56038, Kurume
  - Site Reference ID/Investigator# 55896, Kushiro
  - Site Reference ID/Investigator# 48745, Kyoto
  - Site Reference ID/Investigator# 48746, Kyoto
  - Site Reference ID/Investigator# 48747, Kyoto
  - Site Reference ID/Investigator# 49051, Kyoto
  - Site Reference ID/Investigator# 49053, Kyoto
  - Site Reference ID/Investigator# 49054, Kyoto
  - Site Reference ID/Investigator# 55322, Kyoto
  - Site Reference ID/Investigator# 55577, Kyoto
  - Site Reference ID/Investigator# 55587, Kyoto
  - Site Reference ID/Investigator# 55661, Kyoto
  - Site Reference ID/Investigator# 55718, Kyoto
  - Site Reference ID/Investigator# 55772, Kyoto
  - Site Reference ID/Investigator# 55774, Kyoto
  - Site Reference ID/Investigator# 55775, Kyoto
  - Site Reference ID/Investigator# 55776, Kyoto
  - Site Reference ID/Investigator# 55828, Kyoto
  - Site Reference ID/Investigator# 55829, Kyoto
  - Site Reference ID/Investigator# 60213, Kyoto
  - Site Reference ID/Investigator# 60381, Kyoto
  - Site Reference ID/Investigator# 65102, Kyoto
  - Site Reference ID/Investigator# 65108, Kyoto
  - Site Reference ID/Investigator# 71470, Kyoto
  - Site Reference ID/Investigator# 79893, Kyoto
  - Site Reference ID/Investigator# 94801, Kyoto
  - Site Reference ID/Investigator# 55773, Kyoto, Kyoto
  - Site Reference ID/Investigator# 49044, Machida
  - Site Reference ID/Investigator# 55185, Maebashi
  - Site Reference ID/Investigator# 55697, Maebashi
  - Site Reference ID/Investigator# 55964, Maebashi
  - Site Reference ID/Investigator# 71461, Maebashi
  - Site Reference ID/Investigator# 84198, Marugame
  - Site Reference ID/Investigator# 65147, Matsubushi
  - Site Reference ID/Investigator# 55831, Matsudo
  - Site Reference ID/Investigator# 55832, Matsudo
  - Site Reference ID/Investigator# 55715, Matsue
  - Site Reference ID/Investigator# 48780, Matsumoto
  - Site Reference ID/Investigator# 55159, Matsumoto
  - Site Reference ID/Investigator# 48757, Matsuyama
  - Site Reference ID/Investigator# 48758, Matsuyama
  - Site Reference ID/Investigator# 49071, Matsuyama
  - Site Reference ID/Investigator# 56024, Matsuyama
  - Site Reference ID/Investigator# 60553, Matsuyama
  - Site Reference ID/Investigator# 90417, Matsuyama
  - Site Reference ID/Investigator# 55960, Mibu
  - Site Reference ID/Investigator# 55967, Midori
  - Site Reference ID/Investigator# 49024, Mie
  - Site Reference ID/Investigator# 55632, Mie
  - Site Reference ID/Investigator# 55633, Mie
  - Site Reference ID/Investigator# 55634, Mie
  - Site Reference ID/Investigator# 55635, Mie
  - Site Reference ID/Investigator# 55636, Mie
  - Site Reference ID/Investigator# 55637, Mie
  - Site Reference ID/Investigator# 65119, Mie
  - Site Reference ID/Investigator# 80225, Minato
  - Site Reference ID/Investigator# 49021, Mishima
  - Site Reference ID/Investigator# 55161, Mitaka
  - Site Reference ID/Investigator# 55572, Mitaka
  - Site Reference ID/Investigator# 48656, Mito
  - Site Reference ID/Investigator# 48651, Miyagi
  - Site Reference ID/Investigator# 48653, Miyagi
  - Site Reference ID/Investigator# 48655, Miyagi
  - Site Reference ID/Investigator# 55917, Miyagi
  - Site Reference ID/Investigator# 55918, Miyagi
  - Site Reference ID/Investigator# 55929, Miyagi
  - Site Reference ID/Investigator# 55930, Miyagi
  - Site Reference ID/Investigator# 55931, Miyagi
  - Site Reference ID/Investigator# 55932, Miyagi
  - Site Reference ID/Investigator# 55942, Miyagi
  - Site Reference ID/Investigator# 55943, Miyagi
  - Site Reference ID/Investigator# 60207, Miyagi
  - Site Reference ID/Investigator# 60208, Miyagi
  - Site Reference ID/Investigator# 60379, Miyagi
  - Site Reference ID/Investigator# 60384, Miyagi
  - Site Reference ID/Investigator# 60561, Miyagi
  - Site Reference ID/Investigator# 65150, Miyagi
  - Site Reference ID/Investigator# 67161, Miyagi
  - Site Reference ID/Investigator# 67164, Miyagi
  - Site Reference ID/Investigator# 56055, Miyazaki
  - Site Reference ID/Investigator# 56060, Miyazaki
  - Site Reference ID/Investigator# 56061, Miyazaki
  - Site Reference ID/Investigator# 56063, Miyazaki
  - Site Reference ID/Investigator# 56064, Miyazaki
  - Site Reference ID/Investigator# 80033, Miyazaki
  - Site Reference ID/Investigator# 89837, Monbetsu
  - Site Reference ID/Investigator# 49032, Moriguchi
  - Site Reference ID/Investigator# 48649, Morioka
  - Site Reference ID/Investigator# 89823, Morioka
  - Site Reference ID/Investigator# 89835, Morioka
  - Site Reference ID/Investigator# 90414, Morioka
  - Site Reference ID/Investigator# 89819, Moriya
  - Site Reference ID/Investigator# 55983, Moriyama
  - Site Reference ID/Investigator# 60535, Munakata
  - Site Reference ID/Investigator# 55890, Muroran
  - Site Reference ID/Investigator# 90399, Muroran
  - Site Reference ID/Investigator# 60532, Musashino
  - Site Reference ID/Investigator# 55586, Nagahama
  - Site Reference ID/Investigator# 48685, Nagakute
  - Site Reference ID/Investigator# 55707, Nagano
  - Site Reference ID/Investigator# 55708, Nagano
  - Site Reference ID/Investigator# 55921, Nagano
  - Site Reference ID/Investigator# 55922, Nagano
  - Site Reference ID/Investigator# 55923, Nagano
  - Site Reference ID/Investigator# 60507, Nagano
  - Site Reference ID/Investigator# 60564, Nagano
  - Site Reference ID/Investigator# 48989, Nagaoka
  - Site Reference ID/Investigator# 55582, Nagaoka
  - Site Reference ID/Investigator# 80235, Nagareyama
  - Site Reference ID/Investigator# 48769, Nagasaki
  - Site Reference ID/Investigator# 48770, Nagasaki
  - Site Reference ID/Investigator# 48782, Nagasaki
  - Site Reference ID/Investigator# 49082, Nagasaki
  - Site Reference ID/Investigator# 55866, Nagasaki
  - Site Reference ID/Investigator# 56053, Nagasaki
  - Site Reference ID/Investigator# 56058, Nagasaki
  - Site Reference ID/Investigator# 60211, Nagasaki
  - Site Reference ID/Investigator# 60217, Nagasaki
  - Site Reference ID/Investigator# 60252, Nagasaki
  - Site Reference ID/Investigator# 60266, Nagasaki
  - Site Reference ID/Investigator# 60545, Nagasaki
  - Site Reference ID/Investigator# 65132, Nagasaki
  - Site Reference ID/Investigator# 65133, Nagasaki
  - Site Reference ID/Investigator# 79873, Nagasaki
  - Site Reference ID/Investigator# 94799, Nagasaki
  - Site Reference ID/Investigator# 56011, Nagato
  - Site Reference ID/Investigator# 48683, Nagoya
  - Site Reference ID/Investigator# 48684, Nagoya
  - Site Reference ID/Investigator# 48692, Nagoya
  - Site Reference ID/Investigator# 55608, Nagoya
  - Site Reference ID/Investigator# 55800, Nagoya
  - Site Reference ID/Investigator# 60199, Nagoya
  - Site Reference ID/Investigator# 65107, Nagoya
  - Site Reference ID/Investigator# 71463, Nagoya
  - Site Reference ID/Investigator# 71466, Nagoya
  - Site Reference ID/Investigator# 80223, Nagoya
  - Site Reference ID/Investigator# 84115, Nagoya
  - Site Reference ID/Investigator# 89826, Nagoya
  - Site Reference ID/Investigator# 89828, Nagoya
  - Site Reference ID/Investigator# 94892, Nagoya
  - Site Reference ID/Investigator# 71468, Naha
  - Site Reference ID/Investigator# 55783, Nankoku
  - Site Reference ID/Investigator# 89860, Nankoku
  - Site Reference ID/Investigator# 55680, Nara
  - Site Reference ID/Investigator# 55681, Nara
  - Site Reference ID/Investigator# 55682, Nara
  - Site Reference ID/Investigator# 55683, Nara
  - Site Reference ID/Investigator# 55684, Nara
  - Site Reference ID/Investigator# 94889, Nara
  - Site Reference ID/Investigator# 48669, Narashino
  - Site Reference ID/Investigator# 55701, Narashino
  - Site Reference ID/Investigator# 55788, Narita
  - Site Reference ID/Investigator# 79898, Nasushiobara
  - Site Reference ID/Investigator# 60421, Neyagawa
  - Site Reference ID/Investigator# 48983, Niigata
  - Site Reference ID/Investigator# 48985, Niigata
  - Site Reference ID/Investigator# 48987, Niigata
  - Site Reference ID/Investigator# 48988, Niigata
  - Site Reference ID/Investigator# 48990, Niigata
  - Site Reference ID/Investigator# 49025, Niigata
  - Site Reference ID/Investigator# 55158, Niigata
  - Site Reference ID/Investigator# 55320, Niigata
  - Site Reference ID/Investigator# 55619, Niigata
  - Site Reference ID/Investigator# 55646, Niigata
  - Site Reference ID/Investigator# 55952, Niigata
  - Site Reference ID/Investigator# 55953, Niigata
  - Site Reference ID/Investigator# 65112, Niigata
  - Site Reference ID/Investigator# 49096, Nishihara
  - Site Reference ID/Investigator# 48711, Nishinomiya
  - Site Reference ID/Investigator# 48785, Nishinomiya
  - Site Reference ID/Investigator# 48786, Nishinomiya
  - Site Reference ID/Investigator# 55803, Nishinomiya
  - Site Reference ID/Investigator# 65124, Nishinomiya
  - Site Reference ID/Investigator# 67160, Nishitōkyō
  - Site Reference ID/Investigator# 71471, Nobeoka
  - Site Reference ID/Investigator# 84094, Nomi
  - Site Reference ID/Investigator# 48647, Numakunai
  - Site Reference ID/Investigator# 55842, Numakunai
  - Site Reference ID/Investigator# 55903, Numakunai
  - Site Reference ID/Investigator# 60223, Numakunai
  - Site Reference ID/Investigator# 60249, Numakunai
  - Site Reference ID/Investigator# 60263, Numakunai
  - Site Reference ID/Investigator# 60394, Numakunai
  - Site Reference ID/Investigator# 60538, Numakunai
  - Site Reference ID/Investigator# 68639, Numakunai
  - Site Reference ID/Investigator# 90394, Numata
  - Site Reference ID/Investigator# 48794, Obihiro
  - Site Reference ID/Investigator# 94894, Obihiro
  - Site Reference ID/Investigator# 55187, Odawara
  - Site Reference ID/Investigator# 48749, Okayama
  - Site Reference ID/Investigator# 49055, Okayama
  - Site Reference ID/Investigator# 49056, Okayama
  - Site Reference ID/Investigator# 49059, Okayama
  - Site Reference ID/Investigator# 55984, Okayama
  - Site Reference ID/Investigator# 55988, Okayama
  - Site Reference ID/Investigator# 55989, Okayama
  - Site Reference ID/Investigator# 55990, Okayama
  - Site Reference ID/Investigator# 55991, Okayama
  - Site Reference ID/Investigator# 55992, Okayama
  - Site Reference ID/Investigator# 55995, Okayama
  - Site Reference ID/Investigator# 60390, Okayama
  - Site Reference ID/Investigator# 60527, Okayama
  - Site Reference ID/Investigator# 60529, Okayama
  - Site Reference ID/Investigator# 65127, Okayama
  - Site Reference ID/Investigator# 89822, Okayama
  - Site Reference ID/Investigator# 90398, Okayama
  - Site Reference ID/Investigator# 49097, Okinawa
  - Site Reference ID/Investigator# 55702, Okinawa
  - Site Reference ID/Investigator# 56072, Okinawa
  - Site Reference ID/Investigator# 56074, Okinawa
  - Site Reference ID/Investigator# 56075, Okinawa
  - Site Reference ID/Investigator# 56076, Okinawa
  - Site Reference ID/Investigator# 56078, Okinawa
  - Site Reference ID/Investigator# 56080, Okinawa
  - Site Reference ID/Investigator# 56081, Okinawa
  - Site Reference ID/Investigator# 60255, Okinawa
  - Site Reference ID/Investigator# 60268, Okinawa
  - Site Reference ID/Investigator# 60393, Okinawa
  - Site Reference ID/Investigator# 60420, Okinawa
  - Site Reference ID/Investigator# 60548, Okinawa
  - Site Reference ID/Investigator# 65136, Okinawa
  - Site Reference ID/Investigator# 65137, Okinawa
  - Site Reference ID/Investigator# 79899, Omuta
  - Site Reference ID/Investigator# 79933, Omuta
  - Site Reference ID/Investigator# 89855, Omuta
  - Site Reference ID/Investigator# 48700, Osaka
  - Site Reference ID/Investigator# 48701, Osaka
  - Site Reference ID/Investigator# 48702, Osaka
  - Site Reference ID/Investigator# 48703, Osaka
  - Site Reference ID/Investigator# 48706, Osaka
  - Site Reference ID/Investigator# 49027, Osaka
  - Site Reference ID/Investigator# 49029, Osaka
  - Site Reference ID/Investigator# 49030, Osaka
  - Site Reference ID/Investigator# 49031, Osaka
  - Site Reference ID/Investigator# 49033, Osaka
  - Site Reference ID/Investigator# 49034, Osaka
  - Site Reference ID/Investigator# 49035, Osaka
  - Site Reference ID/Investigator# 49036, Osaka
  - Site Reference ID/Investigator# 49037, Osaka
  - Site Reference ID/Investigator# 55174, Osaka
  - Site Reference ID/Investigator# 55321, Osaka
  - Site Reference ID/Investigator# 55578, Osaka
  - Site Reference ID/Investigator# 55592, Osaka
  - Site Reference ID/Investigator# 55649, Osaka
  - Site Reference ID/Investigator# 55651, Osaka
  - Site Reference ID/Investigator# 55652, Osaka
  - Site Reference ID/Investigator# 55653, Osaka
  - Site Reference ID/Investigator# 55654, Osaka
  - Site Reference ID/Investigator# 55655, Osaka
  - Site Reference ID/Investigator# 55656, Osaka
  - Site Reference ID/Investigator# 55666, Osaka
  - Site Reference ID/Investigator# 55667, Osaka
  - Site Reference ID/Investigator# 55668, Osaka
  - Site Reference ID/Investigator# 55669, Osaka
  - Site Reference ID/Investigator# 55670, Osaka
  - Site Reference ID/Investigator# 55671, Osaka
  - Site Reference ID/Investigator# 55672, Osaka
  - Site Reference ID/Investigator# 55674, Osaka
  - Site Reference ID/Investigator# 55675, Osaka
  - Site Reference ID/Investigator# 55678, Osaka
  - Site Reference ID/Investigator# 55706, Osaka
  - Site Reference ID/Investigator# 55712, Osaka
  - Site Reference ID/Investigator# 55717, Osaka
  - Site Reference ID/Investigator# 60194, Osaka
  - Site Reference ID/Investigator# 60204, Osaka
  - Site Reference ID/Investigator# 60243, Osaka
  - Site Reference ID/Investigator# 60366, Osaka
  - Site Reference ID/Investigator# 60383, Osaka
  - Site Reference ID/Investigator# 60505, Osaka
  - Site Reference ID/Investigator# 60539, Osaka
  - Site Reference ID/Investigator# 60544, Osaka
  - Site Reference ID/Investigator# 60546, Osaka
  - Site Reference ID/Investigator# 60549, Osaka
  - Site Reference ID/Investigator# 60565, Osaka
  - Site Reference ID/Investigator# 65104, Osaka
  - Site Reference ID/Investigator# 65120, Osaka
  - Site Reference ID/Investigator# 65121, Osaka
  - Site Reference ID/Investigator# 67167, Osaka
  - Site Reference ID/Investigator# 67168, Osaka
  - Site Reference ID/Investigator# 79913, Osaka
  - Site Reference ID/Investigator# 89815, Osaka
  - Site Reference ID/Investigator# 90373, Osaka
  - Site Reference ID/Investigator# 60247, Ota-ku, Tokyo
  - Site Reference ID/Investigator# 89853, Ōfunato
  - Site Reference ID/Investigator# 48696, Ōgaki
  - Site Reference ID/Investigator# 48772, Ōita
  - Site Reference ID/Investigator# 49087, Ōita
  - Site Reference ID/Investigator# 49088, Ōita
  - Site Reference ID/Investigator# 49089, Ōita
  - Site Reference ID/Investigator# 49090, Ōita
  - Site Reference ID/Investigator# 49093, Ōita
  - Site Reference ID/Investigator# 55607, Ōita
  - Site Reference ID/Investigator# 56054, Ōita
  - Site Reference ID/Investigator# 56056, Ōita
  - Site Reference ID/Investigator# 56059, Ōita
  - Site Reference ID/Investigator# 56062, Ōita
  - Site Reference ID/Investigator# 60206, Ōita
  - Site Reference ID/Investigator# 60410, Ōita
  - Site Reference ID/Investigator# 67163, Ōita
  - Site Reference ID/Investigator# 68636, Ōita
  - Site Reference ID/Investigator# 89836, Ōita
  - Site Reference ID/Investigator# 55819, Ōme
  - Site Reference ID/Investigator# 48986, Ōsaki
  - Site Reference ID/Investigator# 49057, Ōtsu
  - Site Reference ID/Investigator# 55664, Ōtsu
  - Site Reference ID/Investigator# 55985, Ōtsu
  - Site Reference ID/Investigator# 60522, Ōtsu
  - Site Reference ID/Investigator# 89829, Sabae
  - Site Reference ID/Investigator# 49085, Saga
  - Site Reference ID/Investigator# 56045, Saga
  - Site Reference ID/Investigator# 56046, Saga
  - Site Reference ID/Investigator# 56047, Saga
  - Site Reference ID/Investigator# 56049, Saga
  - Site Reference ID/Investigator# 56050, Saga
  - Site Reference ID/Investigator# 56051, Saga
  - Site Reference ID/Investigator# 60396, Saga
  - Site Reference ID/Investigator# 60503, Saga
  - Site Reference ID/Investigator# 48679, Sagamihara
  - Site Reference ID/Investigator# 55840, Sagamihara
  - Site Reference ID/Investigator# 48673, Saitama
  - Site Reference ID/Investigator# 48674, Saitama
  - Site Reference ID/Investigator# 48676, Saitama
  - Site Reference ID/Investigator# 49014, Saitama
  - Site Reference ID/Investigator# 55323, Saitama
  - Site Reference ID/Investigator# 55606, Saitama
  - Site Reference ID/Investigator# 55833, Saitama
  - Site Reference ID/Investigator# 55834, Saitama
  - Site Reference ID/Investigator# 55835, Saitama
  - Site Reference ID/Investigator# 55836, Saitama
  - Site Reference ID/Investigator# 55838, Saitama
  - Site Reference ID/Investigator# 55839, Saitama
  - Site Reference ID/Investigator# 55845, Saitama
  - Site Reference ID/Investigator# 55846, Saitama
  - Site Reference ID/Investigator# 55847, Saitama
  - Site Reference ID/Investigator# 55848, Saitama
  - Site Reference ID/Investigator# 55849, Saitama
  - Site Reference ID/Investigator# 60197, Saitama
  - Site Reference ID/Investigator# 60419, Saitama
  - Site Reference ID/Investigator# 60526, Saitama
  - Site Reference ID/Investigator# 60534, Saitama
  - Site Reference ID/Investigator# 60541, Saitama
  - Site Reference ID/Investigator# 65118, Saitama
  - Site Reference ID/Investigator# 65149, Saitama
  - Site Reference ID/Investigator# 71472, Saitama
  - Site Reference ID/Investigator# 55308, Sakai
  - Site Reference ID/Investigator# 55676, Sakai
  - Site Reference ID/Investigator# 55677, Sakai
  - Site Reference ID/Investigator# 60512, Sakai
  - Site Reference ID/Investigator# 71469, Sakai
  - Site Reference ID/Investigator# 80221, Sakaidechō
  - Site Reference ID/Investigator# 89861, Sakaidechō
  - Site Reference ID/Investigator# 48993, Saku
  - Site Reference ID/Investigator# 48666, Sakura
  - Site Reference ID/Investigator# 56023, Sanuki
  - Site Reference ID/Investigator# 47382, Sapporo
  - Site Reference ID/Investigator# 48642, Sapporo
  - Site Reference ID/Investigator# 48787, Sapporo
  - Site Reference ID/Investigator# 48789, Sapporo
  - Site Reference ID/Investigator# 48790, Sapporo
  - Site Reference ID/Investigator# 55713, Sapporo
  - Site Reference ID/Investigator# 55868, Sapporo
  - Site Reference ID/Investigator# 55879, Sapporo
  - Site Reference ID/Investigator# 55884, Sapporo
  - Site Reference ID/Investigator# 79956, Sapporo
  - Site Reference ID/Investigator# 89816, Sapporo
  - Site Reference ID/Investigator# 90393, Sapporo
  - Site Reference ID/Investigator# 92733, Sapporo
  - Site Reference ID/Investigator# 92734, Sapporo
  - Site Reference ID/Investigator# 89833, Sasayama
  - Site Reference ID/Investigator# 48771, Sasebo
  - Site Reference ID/Investigator# 48705, Sayama
  - Site Reference ID/Investigator# 48982, Sendai
  - Site Reference ID/Investigator# 55175, Sendai
  - Site Reference ID/Investigator# 55176, Sendai
  - Site Reference ID/Investigator# 55919, Sendai
  - Site Reference ID/Investigator# 79895, Sendai
  - Site Reference ID/Investigator# 89824, Sendai
  - Site Reference ID/Investigator# 60256, Seto
  - Site Reference ID/Investigator# 60516, Setouchi
  - Site Reference ID/Investigator# 55662, Shiga
  - Site Reference ID/Investigator# 55982, Shiga
  - Site Reference ID/Investigator# 55986, Shiga
  - Site Reference ID/Investigator# 55987, Shiga
  - Site Reference ID/Investigator# 60200, Shiga
  - Site Reference ID/Investigator# 60250, Shiga
  - Site Reference ID/Investigator# 60409, Shiga
  - Site Reference ID/Investigator# 94895, Shimada
  - Site Reference ID/Investigator# 55721, Shimane
  - Site Reference ID/Investigator# 60209, Shimane
  - Site Reference ID/Investigator# 60218, Shimane
  - Site Reference ID/Investigator# 65128, Shimane
  - Site Reference ID/Investigator# 65145, Shimane
  - Site Reference ID/Investigator# 89830, Shimizu
  - Site Reference ID/Investigator# 55962, Shimotsuke-shi, Tochigi
  - Site Reference ID/Investigator# 48687, Shizuoka
  - Site Reference ID/Investigator# 49009, Shizuoka
  - Site Reference ID/Investigator# 49012, Shizuoka
  - Site Reference ID/Investigator# 55579, Shizuoka
  - Site Reference ID/Investigator# 55589, Shizuoka
  - Site Reference ID/Investigator# 55609, Shizuoka
  - Site Reference ID/Investigator# 55610, Shizuoka
  - Site Reference ID/Investigator# 55611, Shizuoka
  - Site Reference ID/Investigator# 55881, Shizuoka
  - Site Reference ID/Investigator# 55883, Shizuoka
  - Site Reference ID/Investigator# 60212, Shizuoka
  - Site Reference ID/Investigator# 60374, Shizuoka
  - Site Reference ID/Investigator# 60400, Shizuoka
  - Site Reference ID/Investigator# 60406, Shizuoka
  - Site Reference ID/Investigator# 60418, Shizuoka
  - Site Reference ID/Investigator# 65153, Shizuoka
  - Site Reference ID/Investigator# 89821, Shizuoka
  - Site Reference ID/Investigator# 48753, Shūnan
  - Site Reference ID/Investigator# 55837, Sōka
  - Site Reference ID/Investigator# 89854, Sōka
  - Site Reference ID/Investigator# 55590, Suita
  - Site Reference ID/Investigator# 60365, Suita
  - Site Reference ID/Investigator# 68635, Suwa
  - Site Reference ID/Investigator# 90397, Suzuka
  - Site Reference ID/Investigator# 48698, Tajimi
  - Site Reference ID/Investigator# 48756, Takamatsu
  - Site Reference ID/Investigator# 55173, Takamatsu
  - Site Reference ID/Investigator# 55172, Takarazuka
  - Site Reference ID/Investigator# 89862, Takarazuka
  - Site Reference ID/Investigator# 60372, Takasaki
  - Site Reference ID/Investigator# 90395, Takasaki
  - Site Reference ID/Investigator# 49028, Takatsuki
  - Site Reference ID/Investigator# 55165, Takatsuki
  - Site Reference ID/Investigator# 55648, Takatsuki
  - Site Reference ID/Investigator# 55166, Tenri
  - Site Reference ID/Investigator# 89863, Tenri
  - Site Reference ID/Investigator# 55659, Tochigi
  - Site Reference ID/Investigator# 55961, Tochigi
  - Site Reference ID/Investigator# 60254, Tochigi
  - Site Reference ID/Investigator# 60265, Tochigi
  - Site Reference ID/Investigator# 60562, Tochigi
  - Site Reference ID/Investigator# 67170, Tochigi
  - Site Reference ID/Investigator# 68643, Tochigi
  - Site Reference ID/Investigator# 55628, Toki
  - Site Reference ID/Investigator# 49073, Tokushima
  - Site Reference ID/Investigator# 55314, Tokushima
  - Site Reference ID/Investigator# 55580, Tokushima
  - Site Reference ID/Investigator# 56028, Tokushima
  - Site Reference ID/Investigator# 56029, Tokushima
  - Site Reference ID/Investigator# 71465, Tokushima
  - Site Reference ID/Investigator# 48658, Tokyo
  - Site Reference ID/Investigator# 48659, Tokyo
  - Site Reference ID/Investigator# 48660, Tokyo
  - Site Reference ID/Investigator# 48661, Tokyo
  - Site Reference ID/Investigator# 48662, Tokyo
  - Site Reference ID/Investigator# 48663, Tokyo
  - Site Reference ID/Investigator# 48664, Tokyo
  - Site Reference ID/Investigator# 48665, Tokyo
  - Site Reference ID/Investigator# 48783, Tokyo
  - Site Reference ID/Investigator# 48992, Tokyo
  - Site Reference ID/Investigator# 48996, Tokyo
  - Site Reference ID/Investigator# 48997, Tokyo
  - Site Reference ID/Investigator# 48999, Tokyo
  - Site Reference ID/Investigator# 49003, Tokyo
  - Site Reference ID/Investigator# 49004, Tokyo
  - Site Reference ID/Investigator# 49005, Tokyo
  - Site Reference ID/Investigator# 49007, Tokyo
  - Site Reference ID/Investigator# 55168, Tokyo
  - Site Reference ID/Investigator# 55170, Tokyo
  - Site Reference ID/Investigator# 55191, Tokyo
  - Site Reference ID/Investigator# 55306, Tokyo
  - Site Reference ID/Investigator# 55318, Tokyo
  - Site Reference ID/Investigator# 55575, Tokyo
  - Site Reference ID/Investigator# 55576, Tokyo
  - Site Reference ID/Investigator# 55594, Tokyo
  - Site Reference ID/Investigator# 55595, Tokyo
  - Site Reference ID/Investigator# 55598, Tokyo
  - Site Reference ID/Investigator# 55604, Tokyo
  - Site Reference ID/Investigator# 55695, Tokyo
  - Site Reference ID/Investigator# 55698, Tokyo
  - Site Reference ID/Investigator# 55711, Tokyo
  - Site Reference ID/Investigator# 55714, Tokyo
  - Site Reference ID/Investigator# 55722, Tokyo
  - Site Reference ID/Investigator# 55784, Tokyo
  - Site Reference ID/Investigator# 55786, Tokyo
  - Site Reference ID/Investigator# 55787, Tokyo
  - Site Reference ID/Investigator# 55792, Tokyo
  - Site Reference ID/Investigator# 55795, Tokyo
  - Site Reference ID/Investigator# 55799, Tokyo
  - Site Reference ID/Investigator# 55854, Tokyo
  - Site Reference ID/Investigator# 55867, Tokyo
  - Site Reference ID/Investigator# 55925, Tokyo
  - Site Reference ID/Investigator# 55926, Tokyo
  - Site Reference ID/Investigator# 55927, Tokyo
  - Site Reference ID/Investigator# 55928, Tokyo
  - Site Reference ID/Investigator# 55933, Tokyo
  - Site Reference ID/Investigator# 55934, Tokyo
  - Site Reference ID/Investigator# 55935, Tokyo
  - Site Reference ID/Investigator# 55936, Tokyo
  - Site Reference ID/Investigator# 55937, Tokyo
  - Site Reference ID/Investigator# 55938, Tokyo
  - Site Reference ID/Investigator# 55939, Tokyo
  - Site Reference ID/Investigator# 55940, Tokyo
  - Site Reference ID/Investigator# 55941, Tokyo
  - Site Reference ID/Investigator# 55944, Tokyo
  - Site Reference ID/Investigator# 55945, Tokyo
  - Site Reference ID/Investigator# 60198, Tokyo
  - Site Reference ID/Investigator# 60245, Tokyo
  - Site Reference ID/Investigator# 60370, Tokyo
  - Site Reference ID/Investigator# 60392, Tokyo
  - Site Reference ID/Investigator# 60404, Tokyo
  - Site Reference ID/Investigator# 60417, Tokyo
  - Site Reference ID/Investigator# 60425, Tokyo
  - Site Reference ID/Investigator# 60511, Tokyo
  - Site Reference ID/Investigator# 60514, Tokyo
  - Site Reference ID/Investigator# 60536, Tokyo
  - Site Reference ID/Investigator# 60543, Tokyo
  - Site Reference ID/Investigator# 60547, Tokyo
  - Site Reference ID/Investigator# 65103, Tokyo
  - Site Reference ID/Investigator# 65106, Tokyo
  - Site Reference ID/Investigator# 65113, Tokyo
  - Site Reference ID/Investigator# 65114, Tokyo
  - Site Reference ID/Investigator# 65139, Tokyo
  - Site Reference ID/Investigator# 65142, Tokyo
  - Site Reference ID/Investigator# 68634, Tokyo
  - Site Reference ID/Investigator# 68642, Tokyo
  - Site Reference ID/Investigator# 71462, Tokyo
  - Site Reference ID/Investigator# 71464, Tokyo
  - Site Reference ID/Investigator# 80224, Tokyo
  - Site Reference ID/Investigator# 84096, Tokyo
  - Site Reference ID/Investigator# 89814, Tokyo
  - Site Reference ID/Investigator# 89857, Tokyo
  - Site Reference ID/Investigator# 89874, Tokyo
  - Site Reference ID/Investigator# 48791, Tomakomai
  - Site Reference ID/Investigator# 56073, Tomigusuku
  - Site Reference ID/Investigator# 48742, Tonami
  - Site Reference ID/Investigator# 67166, Toshigi
  - Site Reference ID/Investigator# 48750, Tottori
  - Site Reference ID/Investigator# 55658, Tottori
  - Site Reference ID/Investigator# 55993, Tottori
  - Site Reference ID/Investigator# 55994, Tottori
  - Site Reference ID/Investigator# 55996, Tottori
  - Site Reference ID/Investigator# 55999, Tottori
  - Site Reference ID/Investigator# 48743, Toyama
  - Site Reference ID/Investigator# 49049, Toyama
  - Site Reference ID/Investigator# 55171, Toyama
  - Site Reference ID/Investigator# 55309, Toyama
  - Site Reference ID/Investigator# 55760, Toyama
  - Site Reference ID/Investigator# 55762, Toyama
  - Site Reference ID/Investigator# 60373, Toyama
  - Site Reference ID/Investigator# 60395, Toyama
  - Site Reference ID/Investigator# 60405, Toyama
  - Site Reference ID/Investigator# 49010, Toyoake
  - Site Reference ID/Investigator# 49023, Toyohashi
  - Site Reference ID/Investigator# 94888, Toyokawa
  - Site Reference ID/Investigator# 55754, Toyooka
  - Site Reference ID/Investigator# 89838, Toyooka
  - Site Reference ID/Investigator# 48694, Toyota
  - Site Reference ID/Investigator# 49018, Toyota
  - Site Reference ID/Investigator# 55710, Toyota
  - Site Reference ID/Investigator# 65140, Toyota
  - Site Reference ID/Investigator# 79934, Tōno
  - Site Reference ID/Investigator# 49075, Tōon
  - Site Reference ID/Investigator# 55630, Tsu
  - Site Reference ID/Investigator# 55631, Tsu
  - Site Reference ID/Investigator# 89818, Tsu
  - Site Reference ID/Investigator# 68640, Tsuchiura
  - Site Reference ID/Investigator# 55956, Tsukuba
  - Site Reference ID/Investigator# 60397, Tsuruga
  - Site Reference ID/Investigator# 89859, Tsuruoka
  - Site Reference ID/Investigator# 55777, Uji
  - Site Reference ID/Investigator# 55167, Urayasu
  - Site Reference ID/Investigator# 89825, Usa
  - Site Reference ID/Investigator# 79879, Ushiku
  - Site Reference ID/Investigator# 55830, Utsunomiya
  - Site Reference ID/Investigator# 94890, Utsunomiya
  - Site Reference ID/Investigator# 49045, Wakayama
  - Site Reference ID/Investigator# 49050, Wakayama
  - Site Reference ID/Investigator# 55686, Wakayama
  - Site Reference ID/Investigator# 55687, Wakayama
  - Site Reference ID/Investigator# 55688, Wakayama
  - Site Reference ID/Investigator# 55689, Wakayama
  - Site Reference ID/Investigator# 55690, Wakayama
  - Site Reference ID/Investigator# 55696, Wakayama
  - Site Reference ID/Investigator# 60371, Wakayama
  - Site Reference ID/Investigator# 60391, Wakayama
  - Site Reference ID/Investigator# 60525, Wakayama
  - Site Reference ID/Investigator# 60551, Wakayama
  - Site Reference ID/Investigator# 65123, Wakayama
  - Site Reference ID/Investigator# 67155, Wakayama
  - Site Reference ID/Investigator# 48670, Yachiyo
  - Site Reference ID/Investigator# 55910, Yamagata
  - Site Reference ID/Investigator# 55911, Yamagata
  - Site Reference ID/Investigator# 55915, Yamagata
  - Site Reference ID/Investigator# 55916, Yamagata
  - Site Reference ID/Investigator# 60219, Yamagata
  - Site Reference ID/Investigator# 60267, Yamagata
  - Site Reference ID/Investigator# 60403, Yamagata
  - Site Reference ID/Investigator# 65154, Yamagata
  - Site Reference ID/Investigator# 94803, Yamagata
  - Site Reference ID/Investigator# 48752, Yamaguchi
  - Site Reference ID/Investigator# 48754, Yamaguchi
  - Site Reference ID/Investigator# 49065, Yamaguchi
  - Site Reference ID/Investigator# 49066, Yamaguchi
  - Site Reference ID/Investigator# 49067, Yamaguchi
  - Site Reference ID/Investigator# 55591, Yamaguchi
  - Site Reference ID/Investigator# 55700, Yamaguchi
  - Site Reference ID/Investigator# 56009, Yamaguchi
  - Site Reference ID/Investigator# 56012, Yamaguchi
  - Site Reference ID/Investigator# 56013, Yamaguchi
  - Site Reference ID/Investigator# 56015, Yamaguchi
  - Site Reference ID/Investigator# 60515, Yamaguchi
  - Site Reference ID/Investigator# 94891, Yamatokōriyama
  - Site Reference ID/Investigator# 55679, Yamatotakada
  - Site Reference ID/Investigator# 79896, Yanagawa
  - Site Reference ID/Investigator# 80217, Yanagawa
  - Site Reference ID/Investigator# 60202, Yatomi
  - Site Reference ID/Investigator# 79874, Yatsushiro
  - Site Reference ID/Investigator# 48699, Yokkaichi
  - Site Reference ID/Investigator# 48677, Yokohama
  - Site Reference ID/Investigator# 48678, Yokohama
  - Site Reference ID/Investigator# 55160, Yokohama
  - Site Reference ID/Investigator# 55310, Yokohama
  - Site Reference ID/Investigator# 55852, Yokohama
  - Site Reference ID/Investigator# 55856, Yokohama
  - Site Reference ID/Investigator# 55858, Yokohama
  - Site Reference ID/Investigator# 60399, Yokohama
  - Site Reference ID/Investigator# 60506, Yokohama
  - Site Reference ID/Investigator# 65152, Yokohama
  - Site Reference ID/Investigator# 79954, Yokohama
  - Site Reference ID/Investigator# 89832, Yokohama
  - Site Reference ID/Investigator# 90400, Yokohama
  - Site Reference ID/Investigator# 60424, Yokosuka
  - Site Reference ID/Investigator# 80218, Yokote
  - Site Reference ID/Investigator# 49058, Yonago
  - Site Reference ID/Investigator# 55709, Yonago
  - Site Reference ID/Investigator# 55998, Yonago
  - Site Reference ID/Investigator# 56057, Yufu

REFERENCES:
- [Result] Ogata H, Watanabe M, Matsui T, Hase H, Okayasu M, Tsuchiya T, Shinmura Y, Hibi T. Safety of Adalimumab and Predictors of Adverse Events in 1693 Japanese Patients with Crohn's Disease. J Crohns Colitis. 2016 Sep;10(9):1033-41. doi: 10.1093/ecco-jcc/jjw060. Epub 2016 Mar 9. PMID 26961546
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Humira
Started | 1716
Completed | 1693
Not Completed | 23
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 21

BASELINE CHARACTERISTICS:
Population: Safety analysis set: Excluding 21 patients who were transferred to other institutions during the surveillance period and 2 patients who made no visit after the first administration, 1693 patients were included in the safety analysis set.
Arm/Group | Humira
Number analyzed (Participants) | 1693
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 584
  Male | 1109

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence, which does not necessarily have a causal relationship with treatment. An Adverse Drug Reaction (ADR) is any noxious and undesired reaction related to an experimental drug or experiment. A serious AE (SAE) is an AE that results in death, is life-threatening, results in or prolongs hospitalization, results in congenital anomaly, persistent or significant disability/incapacity, spontaneous or elective abortion, or requires intervention to prevent a serious outcome. AEs were rated for severity as either Mild: transient and easily tolerated; Moderate: causes discomfort and interrupts usual activities; or Severe: causes considerable interference with usual activities, may be incapacitating or life-threatening. AEs related to adalimumab were assessed as being either probably or possibly related by the investigator. An Unexpected ADR is an ADR for which the nature or gravity is not consistent with the applicable product information.
Time Frame: 24 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Humira
Number analyzed (Participants) | 1693
participants
  AEs | 453
  SAEs | 147
  ADRs | 360
  SADRs | 96

2. Primary Outcome: Crohn's Disease Activity Index (CDAI) at Baseline and Week 4
Description: The CDAI is used to evaluate the activity of Crohn's disease. The CDAI is calculated on the basis of a one-week evaluation of 8 items and ranges from 0 to about 600. The 8 items are frequency of liquid or very soft stool, abdominal pain, complications of Crohn's disease (e.g., uveitis, arthritis, fistula, and abscess), abdominal mass, hematocrit, body weight, use of antidiarrheals, and general condition. Low scores indicate low activity of Crohn's disease. In general, CDAI scores below 150 represent remission and scores over 450 represent very severe Crohn's disease.
Time Frame: Baseline, Week 4
Population: Participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Humira
Number analyzed (Participants) | 1017
scores on a scale
  Baseline (n=1017) | 204.3 (105.7)
  Week 4 (n=912) | 142.9 (90.4)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Paired t-test using observed cases at Baseline and Week 4

3. Secondary Outcome: Improvement Rating by Investigator at Week 24
Description: Overall response rating, according to investigator's subjective clinical opinion. The level of improvement (markedly improved, improved, not improved, or not assessable) was categorized by comparing clinical condition at week 24 or at discontinuation with baseline condition.
Time Frame: Week 24
Measure: Number; unit: percentage of participants
Arm/Group | Humira
Number analyzed (Participants) | 1619
percentage of participants
  Percentage of Participants Markedly improved | 20.6
  Percentage of Participants Improved | 55.3
  Percentage of Participants Not Improved | 17.2
  Percentage of Participants Not Assessable | 7.0

4. Primary Outcome: Crohn's Disease Activity Index (CDAI) at Baseline and Week 8
Description: as for outcome 2
Time Frame: Baseline, Week 8
Population: Participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Humira
Number analyzed (Participants) | 1017
scores on a scale
  Baseline (n=1017) | 204.3 (105.7)
  Week 8 (n=818) | 142.7 (93.8)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Paired t-test using observed values at Baseline and Week 8

5. Primary Outcome: Crohn's Disease Activity Index (CDAI) at Baseline and Week 24
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: Participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Humira
Number analyzed (Participants) | 1017
scores on a scale
  Baseline (n=1017) | 204.3 (105.7)
  Week 24 (n=982) | 149.1 (100.9)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Paired t-test using observed values at Baseline and Week 24

6. Secondary Outcome: Remission Rate at Week 4, Week 8, and Week 24
Description: The remission rate for each evaluation timepoint (Weeks 4, 8, and 24) was calculated as the number of participants that had CDAI < 150 divided by the number of participants at Baseline that had CDAI scores ≥ 150.
Time Frame: Baseline, Week 4, Week 8, and Week 24
Population: Participants with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Humira
Number analyzed (Participants) | 1017
percentage of participants
  Week 4 (284/607) | 46.8
  Week 8 (260/542) | 48.0
  Week 24 (304/649) | 46.8

ADVERSE EVENTS:
Time Frame: 24 weeks.
Arm/Group | Humira
Serious Adverse Events (participants affected / at risk) | 147/1693
Other Adverse Events (participants affected / at risk) | 177/1693
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (N=1693)
Abdominal wall abscess (Infections and infestations) | 1
Abscess intestinal (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cholangitis suppurative (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Pelvic abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 6
Postoperative wound infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Tonsillitis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vestibular neuronitis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 7
Salpingo-oophoritis (Infections and infestations) | 1
Intestinal fistula infection (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Lung infection pseudomonal (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Abdominal abscess (Infections and infestations) | 4
Pneumonia bacterial (Infections and infestations) | 1
Chlamydial infection (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Enterocolitis viral (Infections and infestations) | 1
Herpes ophthalmic (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Infectious peritonitis (Infections and infestations) | 3
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Panic disorder (Psychiatric disorders) | 1
Adjustment disorder (Psychiatric disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cranial nerve palsies multiple (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Mononeuropathy multiplex (Nervous system disorders) | 1
Vasculitis cerebral (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiovascular disorder (Cardiac disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Anal stenosis (Gastrointestinal disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal stenosis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
IIleal stenosis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 4
Intestinal obstruction (Gastrointestinal disorders) | 9
Intestinal perforation (Gastrointestinal disorders) | 1
Intestinal stenosis (Gastrointestinal disorders) | 5
Large intestine perforation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 4
Pancreatitis acute (Gastrointestinal disorders) | 1
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 7
Enterocutaneous fistula (Gastrointestinal disorders) | 1
Anorectal varices haemorrhage (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal haemorrhage (Renal and urinary disorders) | 1
Chest discomfort (General disorders) | 1
Malaise (General disorders) | 1
Multi-organ failure (General disorders) | 1
Pyrexia (General disorders) | 4
Sudden death (General disorders) | 1
Blood creatine phosphokinase increased (Investigations) | 2
Blood pressure increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Administration related reaction (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (N=1693)
Bronchitis (Infections and infestations) | 10
Influenza (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 30
Pharyngitis (Infections and infestations) | 13
Anaemia (Blood and lymphatic system disorders) | 8
Headache (Nervous system disorders) | 9
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 13
Nausea (Gastrointestinal disorders) | 9
Hepatic function abnormal (Hepatobiliary disorders) | 9
Liver disorder (Hepatobiliary disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 24
Injection site erythema (General disorders) | 11
Injection site reactions (General disorders) | 24
Malaise (General disorders) | 9
Pyrexia (General disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.